CLINICAL TRIAL: NCT02182375
Title: An Open Label Fixed Sequence Phase I Study to Investigate the Effect of BI 201335 Mediated UGT1A1 Inhibition on the Multiple Oral Dose Pharmacokinetics of Raltegravir (Isentress®) in Healthy Male and Female Volunteers
Brief Title: Effect of BI 201335 Mediated UGT1A1 (Uridine-diphosphate-glucuronosyltransferases) Inhibition in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1220.9
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Raltegravir Potassium

ARMS (1):
- BI 201335 NA (Experimental): 400 mg raltegravir (bid) from day 1-14 and once on day 15;
  240 mg BI 201335 NA (bid) from day 7-14 with a loading dose of 480 mg in the morning of day 6 and once on day 15
  Interventions: Drug: BI 201335 NA; Drug: Raltegravir

INTERVENTIONS:
Drug: BI 201335 NA
Drug: Raltegravir

SUMMARY:
Study to investigate the effect of UGT1A1 inhibition by single and multiple oral doses of BI 201335 on the single and multiple oral dose pharmacokinetics of raltegravir and to investigate safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Age ranging ≥ 21 and ≤ 50 years
* Body mass index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2
* Willing to complete all study-related activities including genotyping
* Volunteers give their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG (Electrocardiogram)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, clinically relevant electrolyte disturbances
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of photosensitivity or recurrent rash
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or clinically relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study (with the exception of hormonal contraceptives)
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the trial or during the trial
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (> 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range if indicative of underlying disease or poor health
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to treatment medication and/or related drugs of these classes
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTcF, or QTcB interval >450 ms)
* Vulnerable subjects (that is persons kept in detention)
* The subject is not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
* For Female Subjects:

  * Pregnancy
  * Positive pregnancy test
  * Lactation period
  * No adequate contraception: females participating in the study must be either (1) of non-childbearing potential (e.g. surgically sterilized or postmenopausal with no menstrual bleeding for at least 2 years prior the study), or (2) using one of the following contraceptive methods plus condom during the course of the study and up to one month (i.e. one complete menstrual cycle) after the last administration of the study drug (whichever is longer): implants of levonorgestrel or injectable progestogen, oral contraceptive - combined or progestogen only, intrauterine device (IUD)- any IUD with published data showing that the lowest expected failure rate is less than 1% per year (not all IUDs meet this criteria)
* For Male Subjects:

  * No adequate contraception: (1) surgically sterilized or (2) or use a condom plus another form of contraception (e.g. spermicide, IUD, birth control pills taken by female partner, diaphragm with spermicide). Male subjects must not father a child from administration of the first dose and up to 3 months after the last dose of study medication

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Steady-state Cmax,ss (maximum measured concentration) of raltegravir and raltegravir glucuronide | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 5, 7 and 15
Steady-state AUC0-12h,ss (Area under the concentration-time curve) of raltegravir and raltegravir glucuronide | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 5, 7 and 15
C12h,ss of raltegravir and raltegravir glucuronide | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 5, 7 and 15

SECONDARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline and within 7-14 days after last treatment
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | Baseline and days 1, 5, 6, 7, 15 and within 7-14 days after last treatment
Number of patients with adverse events | up to 7 - 14 days after last treatment
Number of patients with abnormal findings in 12-lead ECG (electrocardiogram) | Baseline, days 1, 5, 6, 7, 15 and within 7-14 days after last treatment
Number of patients with abnormal changes in laboratory tests (hematology, clinical chemistry, urine analysis) | Baseline, days 1, 2, 5, 6, 7, 8, 10, 12, 14, 15, 16 and within 7-14 days after last treatment
Assessment of tolerability by investigator on a 4-point scale | within 7-14 days after last treatment
Cmax,ss of BI 201335 ZW | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 7 and 15
C12h,ss of BI 201335 ZW | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 7 and 15
AUC0-12,ss of BI 201335 ZW | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 7 and 15
tmax,ss (Time from dosing to the maximum measured concentration) of BI 201335 ZW | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 7 and 15
CL/F0-12,ss (Total apparent clearance) of BI 201335 ZW | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 7 and 15
V/F0-12,ss (Apparent volume of distribution) of BI 201335 ZW | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 7 and 15
tmax,ss of raltegravir and raltegravir glucuronide | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 5, 7 and 15
CL/F0-12,ss of raltegravir | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 5, 7 and 15
V/F0-12,ss of raltegravir | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 5, 7 and 15
t1/2 of raltegravir and raltegravir glucuronide | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose on day 5, 7 and 15
Ae (Amount of analyte eliminated in urine) of raltegravir and raltegravir glucuronide | pre-dose and 0-4, 4-8, 8-12 hours post-dose on day 5, 7, 15
CLR (Renal clearance) of raltegravir and raltegravir glucuronide | pre-dose and 0-4, 4-8, 8-12 hours post-dose on day 5, 7, 15
fe (Fraction of analyte eliminated in urine) of raltegravir and raltegravir glucuronide | pre-dose and 0-4, 4-8, 8-12 hours post-dose on day 5, 7, 15